CLINICAL TRIAL: NCT00907374
Title: Early Nephropathy Study in Diabetes With Inhibitory Renin-Angiotensin-Aldosterone System Therapy (END-IT)
Brief Title: Low Dose Versus Aggressive Inhibition of the Renin-Angiotensin-Aldosterone (RAS) to Treat Microalbuminuria
Acronym: END-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Responsible Party: Principal Investigator, Mayer Davidson, Professor of Medicine, Charles Drew University of Medicine and Science
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB# 04-09-772; U54RR014616 (NIH)
Record Dates: First submitted 2009-05-21; First posted 2009-05-22 (Estimated); Results first posted 2012-03-30 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Microalbuminuria
Keywords: Microalbuminuria; Carotid intima media thickness; Endothelial dysfunction; Renin angiotensin system; Diabetic nephropathy
MeSH Terms: conditions — Diabetic Nephropathies | interventions — benazepril; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low dose inhibition of RAS (Active Comparator): Standard low dose inhibition of the RAS with 10 mg of benazepril orally daily to treat microalbuminuria
  Interventions: Drug: benazepril
- Agressive inhibition of the RAS (Experimental): 40-80 mg benazepril plus 25-100 mg losartan both orally once or twice daily
  Interventions: Drug: benazepril

INTERVENTIONS:
Drug: benazepril — benazepril 10 mg orally once daily
  Other Names: Lotensin
  Arms: Low dose inhibition of RAS
Drug: benazepril — 40-80 mg benazepril plus 25-100 mg losartan orally once or twice daily
  Other Names: Lotensin; Cozaar
  Arms: Agressive inhibition of the RAS

SUMMARY:
The objective of the study is to assess the effect of standard versus aggressive inhibition of the renin-angiotensin system (RAS)in type 2 diabetic patients with microalbuminuria (MA) on; a)progression of microalbuminuria, b)estimated glomerular filtration rate (eGFR), c)endothelial dysfunction (measured by post-hyperemia arterial tonometry) and d)the slowing of the progression of atherosclerotic disease (measured by carotid intima media thickness [CIMT]).

DETAILED DESCRIPTION:
Diabetic patients with confirmed MA (50-300 mg albumin per g creatinine) on a morning spot urine sample were entered into a one to three month run-in phase before randomization. (50 mg/g was used as the lower limit to allow room for improvement to reach normal.) Since hypertension and uncontrolled hyperglycemia will cause MA, blood pressure (BP) and hemoglobin A1c (AIC) levels were reduced to <130/80 mm Hg and <8.0%, respectively, during this period. All patients had been on various doses of an angiotensin converting enzyme inhibitor (ACE-I) which were reduced to 10 mg benazepril and BP controlled with other classes of anti-hypertensive drugs (except for angiotensin receptor blockers [ARB's]). Glycemia was treated with intensification of their current therapy. MA and BP were measured monthly.

When goal levels of BP and AIC were achieved and MA was still present, patients were randomized to either low dose RAS inhibition (10 mg benazepril) (Standard) or aggressive inhibition of the RAS (Aggressive). MA continued to be measured monthly and the progressive increase in doses of an ACE-I and an ARB was as follows. Benazepril (the ACE-I) - 10 mg to 20 mg to 40 mg to adding losartan (the ARB) -25 mg to 50 mg to 100 mg to increasing benazepril to 80 mg with the goal of returning albumin excretion to normal. Other classes of drugs were reduced as necessary to keep systolic BP > 100 mm Hg. Serum creatinine and potassium[K+] were measured monthly, AIC levels every 3 months and CIMT by ultrasound and endothelial function by post hyperemia and nitroglycerine (NTG) - induced peripheral artery tonometry (PAT) via finger plethysmography every six months.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age 18-70
* Subjects with diabetic renal disease as defined by spot urine albumin - creatinine ratio 30-300mg/g and estimated glomerular filtration rate of >60 ml/min

Exclusion Criteria:

* Intake of non-steroidal anti-inflammatory agents (NSAIDs) more than 15 days/month, excluding aspirin.
* Inability to discontinue NSAIDs or aspirin for 5 days prior to GFR measurement.
* History of severe adverse reaction to any of the randomized drugs required for use in the protocol or contraindication of their use.
* Participation in another intervention study.
* Pregnancy or likelihood of becoming pregnant during the study period; lactation
* Clinical and laboratory evidence of any renal disease other than diabetic nephropathy.
* History of drug abuse in the past 2 years, including narcotics, cocaine or alcohol (> 21 drinks per week). Serious systemic disease that might influence survival or the course of renal disease. (Chronic oral steroid therapy is exclusion, but steroid-containing nasal sprays are not. Inactive sarcoidosis is not an exclusion).
* History of malignant or accelerated hypertension within 6 months prior to study entry; previous chronic peritoneal or hemodialysis or renal transplantation. Known secondary causes of hypertension. Spot urine albumin - creatinine ratio exceeding 300 (mg/g)
* Serum potassium level > 5.5 mEq/L for those not on ACE inhibitors during Baseline, or serum potassium level > 5.9 mEq/L for those on ACE inhibitors during Baseline.

Leukopenia < 2,500/mm3 at screening and confirmed at the end of Baseline.

* Doubt that the participant will be able to adhere to medications or comply with the protocol visit schedule
* Arm Circumference > 52 cm, which precludes measuring blood pressure with the "thigh" blood pressure cuff. Arm length such that if the cuff circumference extended into the antecubital space so that the cuff interfered with placement of the stethoscope over the brachial artery for blood pressure measurement
* Clinical evidence of lead intoxication. Clinical evidence of congestive heart failure, current or within the preceding six months. Ejection fraction below 35% measured by any method. Heart block greater than first degree or any other arrhythmia that contraindicated the use of any of the primary BP drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2005-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naureen Taureen, MD, Principal Investigator — Charles Drew University; Mayer B. Davidson, MD, Study Director — Charles Drew University
Locations (1):
- Charles Drew University, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 46 patients were enrolled and entered the run-in but 19 were not randomized
Groups:
- Low Dose Inhibition of RAS: 10 mg benazepril plus other anti-hypertensive agents to treat elevated BP
- Agressive Inhibition of the RAS: 40-80 mg benazepril plus 25-100 mg losartan both p.o. 1-2X per day
Period: Overall Study
Arm/Group | Low Dose Inhibition of RAS | Agressive Inhibition of the RAS
Started | 14 | 13
Completed | 12 | 11
Not Completed | 2 | 2
Not completed — Noncompliant w/study protocol at <3 mos | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Inhibition of RAS | Agressive Inhibition of the RAS | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 27
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 54.4 (6.7) | 51.6 (5.9) | 53.0 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Microalbuminuria Reported as Urinary Albumin:Creatinine Ratio
Description: Average of ratio for all participants during the 3-36 months of the study
Time Frame: 3 to 36 months
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Low Dose Inhibition of RAS | Agressive Inhibition of the RAS
Number analyzed (Participants) | 12 | 11
Ratio | 256.1 (652.3) | 376.2 (404.2)

2. Secondary Outcome: Estimated Glomerular Filtration Rate
Description: This is an average for all participants during the 3-36 month study period
Time Frame: 3 to 36 months
Population: Completers
Measure: Mean (Standard Deviation); unit: ml/min/1.73 meters squared
Arm/Group | Low Dose Inhibition of RAS | Agressive Inhibition of the RAS
Number analyzed (Participants) | 12 | 11
ml/min/1.73 meters squared | 108.7 (21.6) | 100.5 (33.7)

3. Secondary Outcome: Carotid Artery Intima Thickness
Description: Thickness of intima of right carotid artery; average of all particpants from 6-36 months of study
Time Frame: 6 to 36 months
Population: Completers
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Low Dose Inhibition of RAS | Agressive Inhibition of the RAS
Number analyzed (Participants) | 12 | 11
mm | 0.74 (0.09) | 0.72 (0.17)

4. Secondary Outcome: Endothelial Dysfunction
Description: Post hyperemia increase in blood flow - fold increase from before and after occluding BP; values are mean of all participants in 6-36 months of study period.
Time Frame: 6 to 36 months
Population: complerters
Measure: Mean (Standard Deviation); unit: Fold increase
Arm/Group | Low Dose Inhibition of RAS | Agressive Inhibition of the RAS
Number analyzed (Participants) | 12 | 11
Fold increase | 2.2 (0.5) | 2.0 (0.7)

ADVERSE EVENTS:
Arm/Group | Low Dose Inhibition of RAS | Agressive Inhibition of the RAS
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 2/13
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Inhibition of RAS (N=14) | Agressive Inhibition of the RAS (N=13)
Systolic BP <100 mm Hg (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No